CLINICAL TRIAL: NCT03615027
Title: Dementia-specific Intervention of Advance Care Planning
Acronym: ADIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Francesca Bosisio, Research assistant, University of Lausanne Hospitals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-00785
Record Dates: First submitted 2018-06-21; First posted 2018-08-03 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: This clinical trial has a sigle arm: all the dyads will go through the four visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): see detailed description
  Interventions: Behavioral: Dementia-specific advance care planning

INTERVENTIONS:
Behavioral: Dementia-specific advance care planning — see detailed description

SUMMARY:
This is a pilot study that aims to create a dementia-specific intervention of advance care planning (ACP) and test its feasibility and acceptance with min 20 max 30 patient-relative dyads.

The intervention is adapted from the Multiprofessional advance care planning and shared decision-making for end of life care (MAPS) Trials 1 and 2 made at the Zurich University Hospital.

The study design is longitudinal (historic): all the dyads will be asked to go through the process (4 visits, see 9.3 Procedures at each visit).

DETAILED DESCRIPTION:
Study background and aims:

Advance care planning (ACP) is a structured communication process between an individual, his family, and his healthcare agent (if existing), facilitated by a healthcare provider. The aim is to identify the personal values of the individual, reflect on the meanings and consequences of anticipated illness scenarios, define goals and preferences of care for these situations, issue appropriate documents and legal instruments that will help direct future healthcare decisions, and review these steps at adequate intervals. ACP emphasizes communication in anticipation of a future deterioration of a person's health. Even though dementia entails the loss of decision-making capacity, advance care planning is yet to become widespread. This study aims to close the gap and create a dementia-specific ACP intervention that:

* Support patient autonomy through advance care planning
* Improve participants' satisfaction and perceived control;
* Increase planning decisions and surrogate's knowledge of patients' preferences and values.

Procedure and measure:

Pre-intervention assessment (Visit 1):

If the patient and her/his relative have both consented to the study, the PI will ask the patient and her/his relative to fil out psychometric scales: Hospital anxiety and depression scale (HADS), Decisional conflict scale, Personal autonomy scale and Zarit Burden Inventory. Then, the PI will realize a semi-structured interview on patient's val-ues and treatment preferences and caregiver's knowledge of patient's preferences and care planning decisions that have already been made. Participants will also be asked to hand out a copy of any pre-existing advance directives or other advance care planning document.

Intervention (Visit 2):

In the intervention this first conversation (45-90 min) with a specifically trained ACP facilitator aims to explain the goal and content of ACP and prompt the patient to reflect upon his/her values and preferences for healthcare and discuss them with his/her caregiver. In addition, the written decision aids will be explained and provided to the patient/caregiver to be read at home. At the end of the meeting, the facilitator will ask to set up the second meeting.

Intervention (Visit 3):

The second conversation of the ACP facilitator with the patient and her/his caregiver aims to help the patient to specify her/his preferences and trans-late them into actionable documentation. The discussions also aim to empower the caregiver to make sure that these decisions are respected.

Post-intervention assessment (Visit 4):

The PI will start the meeting with a semi-structured interview (30-45 min) on the dyad's subjective experience with the intervention, positive and nega-tive effects, and challenges and suggestions to modify the intervention. Participants will also be asked to hand over copies of ACP documents produced during the intervention or after it in order to be analysed. After the interview, the PI will ask the patient and her/his relative to fill in psychometric scales: Hospital anxiety and depression scale (HADS), Decisional conflict scale, Personal autonomy scale and Zarit Burden Inventory.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 65 years
* Having been diagnosed with an early-stage dementia of Alzheimer's disease aetiology or mixed Alzheimer-vascular aetiology (Montreal cognitive assessement (MoCA) > 20 and Clinical dementia rating (CDR) < 1.5);
* Having been informed about the diagnosis by their treating physician and that are regularly followed by him/her;
* Patient that show interest in advance care planning or advance directives;
* Patients with psychiatric disorders can be included if their psychiatric symptoms are controlled and under the supervision of their psychiatrist at the Unit of psychogeriatric care;
* Retaining full decision-making capacity according to the MoCA > 20 or the clinical judgement a physician or psychologist. During the study, the PI and the facilitators will monitor patient's decision-making capacity clinically;
* Having the necessary French language competencies to engage in conversations;
* Having a close family caregiver over 18 years old, who is informed about the patient's diagnosis, possesses the before mentioned cognitive and communication skills, and is willingly to participate to this pilot intervention;
* Informed Consent for both members of the dyad as documented by signature;

Exclusion Criteria:

* Patients that have a dementia associated with fronto-temporal lobe degeneration;
* Patients that have mild cognitive impairments (MCI);
* Patients that have moderate to severe cognitive disorders, anosognosia or else, assessed clinically or through scales or based on in-person screening, that suggest decision-making capacity may be impaired;
* The patient or her/his caregiver decide to withdraw from the study;
* Enrolment of the investigator, his/her family members, employees and other dependent persons.
* Patients that have a dementia associated with fronto-temporal lobe degeneration;
* Patients that have MCI;
* Patients that have moderate to severe cognitive disorders, anosognosia or else, assessed clinically or through scales or based on in-person screening, that suggest decision-making capacity may be impaired;
* The patient or her/his caregiver decide to withdraw from the study;
* Enrolment of the investigator, his/her family members, employees and other dependent persons.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08-03 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in participants' anxiety and depression levels | Visit 1 and V4 (=V1 + 4-6 weeks)
  Changes in participants' anxiety and depression levels measured with the Hospital Anxiety and Depression scale before (V1) and after (V4) the intervention. The Hospital Anxiety and Depression Scale (HADS) allow the participant to assess her/his mood according to 24 items. Individual's anxiety and depression levels are calculated by summing the score obtained at the eponym subscales, 0 being no anxiety or depression and 21 high anxiety or depression.
Change in participants' decisional conflict level | Visit 1 and V4 (=V1 + 4-6 weeks)
  Changes in participants' decisional conflict levels measured with the Decisional conflict scale before (V1) and after (V4) the intervention. The decisional conflict scale allow to participant to assess her/his ambivalence towards a specific treatment decision by choosing on a Lickert scale whether s/he strongly agrees (0 points), agrees (1 point), neither agrees nor disagrees (2 points), disagrees (3 points), or strongly disagrees (4 points) with a list of sentences. Scores are then summed, divided by 16 and multiplied by 25. Scores range from 0 (no decisional conflict) to 100 (extremely high decisional conflict).
Change in proxies' perception of the burden | Visit 1 and V4 (=V1 + 4-6 weeks)
  Changes in relative's perceptions of the burden measured with the Zarit Burden Inventory before (V1) and after (V4) the intervention. The Zarit Burden Inventory assesses relative's perceived burden of taking care of a sick and/or dependent loved one. Relatives have to answer to indicate if they experienced 22 different situations or feelings never (1 point), rarely (2 points), sometimes (3 points), quite frequently (4 points), or nearly always (5 points). Points at each item are summed: scores range from 22 (low perceived burden) to 110 (high perceived burden).
Changes in patients' psychological autonomy and perceived control | Visit 1 and V4 (=V1 + 4-6 weeks)
  Changes in perceptions of patient's personal autonomy measured with the Psychological Autonomy Inventory before (V1) and after (V4) the intervention. The Psychological Autonomy Inventory allows the patient to indicate on a scale from 1 to 5 (1 being never and 5 all the time) how s/he feels autonomous in different aspects of life. Scores at the subscale of decisional control (items 3, 7, 10, 12, 14, 15, 16, 18, 19, 20, 25, 26, 27, and 28) are summed. Items at the subscale of behavioral control (items 1, 2, 4, 5, 6, 8, 9, 11, 13, 17, 21, 22, 23, and 24) are summed. A score of 14 means low decisional or behavioral control, a score of 70 means high decisional or behavioral control.
Participants' satisfaction with the intervention | Visit 1 and V4 (=V1 + 4-6 weeks)
  Semi-structured interview at V4 explores dyad's experience with the intervention, whether advance decisions were documented during or after the intervention and how, and comments and suggestions to improve the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Lausanne University Hospital, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared outside of the research group or for other studies

REFERENCES:
- [Derived] Bosisio F, Sterie AC, Rubli Truchard E, Jox RJ. Implementing advance care planning in early dementia care: results and insights from a pilot interventional trial. BMC Geriatr. 2021 Oct 19;21(1):573. doi: 10.1186/s12877-021-02529-8. PMID 34666711